CLINICAL TRIAL: NCT07008807
Title: The Facial Muscular Activity: A Paradigm for Understanding Facial Asymmetry, A Prospective Correlation Study
Brief Title: The Facial Muscular Activity: A Paradigm for Understanding Facial Asymmetry
Status: Not yet recruiting | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed E. Ali, Lecturer of Physical Therapy for surgery, South Valley University
Other Study IDs: SREC.PT.SUE(7)325
Record Dates: First submitted 2025-05-20; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Facial Asymmetry
MeSH Terms: conditions — Facial Asymmetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: people with facial asymmetry
- Group B: control group of healthy normal people

SUMMARY:
Facial asymmetry, the degree to which the two sides of the face differ in size, shape, or the arrangement of features, is a near-universal human characteristic. The intricate network of facial muscles plays a crucial role in both the static structure and the dynamic expressions of the face. The continuous pull and action of facial muscles can influence the development and positioning of underlying soft tissues and even, over extended periods, potentially impact skeletal structures.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with noticeable facial asymmetry
* Age > 16 years
* General good health
* Absence of specific neurological conditions affecting facial muscles.
* Absence of congenital facial disorders that might cause facial asymmetry, like hemifacial microsomia and cleft lip and palate syndromes.

Exclusion Criteria:

* History of facial trauma or surgery
* Diagnosed Neuromuscular Disorders
* Active facial infections.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Presenting with noticeable facial asymmetry.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Facial Electromyography (EMG) | Day 1
Facial Asymmetry Measurement | Day 1
  assesses differences between the two sides of the face using various techniques, both two-dimensional (2D) and three-dimensional (3D)

SECONDARY OUTCOMES:
Demographic and Clinical Data | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- orthodontic outpatient clinic, and students at Faculty of Dentistry, Alsalam University, Egypt, Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 4. Kowner, R. (1996). Facial asymmetry and attractiveness judgment in Western and Japanese cultures. Journal of Social Behavior and Personality, 11(2), 301-314.
- [Background] Ferrario VF, Dellavia C, Tartaglia GM, Turci M, Sforza C. Soft tissue facial morphology in obese adolescents: a three-dimensional noninvasive assessment. Angle Orthod. 2004 Feb;74(1):37-42. doi: 10.1043/0003-3219(2004)0742.0.CO;2. PMID 15038489